CLINICAL TRIAL: NCT01365442
Title: Pilot Introduction of the Modified Bivalent Killed Whole Cell Oral Cholera Vaccine in Orissa
Brief Title: Pilot Introduction of Oral Cholera Vaccine in Orissa, India
Status: Completed | Type: Observational
Sponsor: International Vaccine Institute (Other)
Collaborators: Department of Health and Family Welfare, Orissa (Other); Indian Council of Medical Research (Other Government); National Institute of Cholera and Enteric Diseases, India (Other); Shantha Biotechnics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-WC-03
Record Dates: First submitted 2010-03-10; First posted 2011-06-03 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Cholera
Keywords: Cholera; Vaccination; Oral cholera vaccine; Mass vaccination; Oral whole cell cholera vaccine
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Observational Model: Ecologic or Community
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consenting, eligible participants: All consenting eligible participants in the study area will receive the oral cholera vaccine

SUMMARY:
The purpose of this study is to provide evidence for policymakers and key opinion leaders on the pilot implementation of cholera vaccination using the newly licensed Oral Cholera Vaccine (OCV) in India. The pilot introduction will provide the evidence for the feasibility, costs and population acceptance of large-scale cholera vaccination using the Indian vaccine (using vaccination coverage rates and other measures).

DETAILED DESCRIPTION:
Severe diarrhoeal disease caused by Vibrio cholerae O1 and O139 has long been an important cause of mortality and morbidity in India. The availability and recent licensure of the modified bivalent killed whole cell OCV in India provides hope that the disease may be controlled in areas where the disease is a problem. On April 10, 2009, a meeting was organized by the Indian Council of Medical Research (ICMR), the Department of Biotechnology and the IVI. The recommendations from the meeting are as follows:

* As the modified WC vaccine is safe, effective, and cost-effective, it was suggested that the National Technical Advisory Group on Immunization (NTAGI) should consider recommending introduction of the vaccine in public health programs targeted to appropriate populations in India.
* Vaccination should be initiated in selected highly endemic and/or slum areas such as known areas in West Bengal or Orissa. The pilot vaccination programs will be monitored and evaluated. Further expansion to other areas and wider policy changes will be made in a step-by-step fashion based on the pilot programs. Logistical and operational issues need to be defined.

The aim of the study is to conduct a pilot introduction of the modified killed oral cholera vaccine in a public health setting in a population of ~50,000 before implementing in a larger scale.

Primary objective:

To determine the feasibility, acceptability and costs associated with pilot introduction of the modified killed whole cell oral cholera vaccine in India when given in a public health setting.

Secondary objective:

To identify challenges to mass oral cholera vaccine implementation.

ELIGIBILITY:
Inclusion Criteria:

* aged 12 months and older
* non-pregnant

Exclusion Criteria:

* age less than 12 months
* pregnant
* too ill/old to get out of bed

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted in ~100 selected villages with approximate population of 50,000 in Satyabadi block of Puri district, Orissa
Sampling Method: Non-Probability Sample
Enrollment: 31552 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility | The numerator (number of people who received the vaccine doses within the target population) will be counted during the 30 days following the last dose of vaccination.
  Feasibility will be determined by the vaccine coverage (%), defined as the number of subjects who received the vaccine doses divided by the number of subjects who are targeted for mass vaccination.

SECONDARY OUTCOMES:
Assessment of acceptability and costs of vaccination program | For a thirty days starting from the 30 days following the last dose of vaccination
  Costs of vaccination program will be defined as the sum of the cost items required for social mobilization, mass vaccination, and post-vaccination actiities. This includes 1) vaccine price, 2) shipment and insurance costs, 3) personnel(FTEs), 4) supplies including coldboxes and vaccine carriers, 5) transportation.
  Acceptability will be evaluated by
  1. vaccine coverage rate
  2. survey results which will be qualtitaviely and quantitatively summarized by the sociobehavioral scientists based on in-person interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Shantanu K Kar, MD, Principal Investigator — Director, Regional Medical Research Center, Bhubaneswar, Orissa, India
Locations (1):
- Regional Medical Research Center, Chandrashekharpur, Bhubaneswar, Odisha, India